CLINICAL TRIAL: NCT02132754
Title: Phase 1 Trial of Single Agent MK-4166 and MK-4166 in Combination With Pembrolizumab in Subjects With Advanced Malignancies
Brief Title: Study of MK-4166 and MK-4166 in Combination With Pembrolizumab (MK-3475) in Participants With Advanced Solid Tumors (MK-4166-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4166-001; MK-4166-001 (Other: Merck)
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Results first posted 2020-07-31 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — MK-4166; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (34):
- MK-4166 0.0015 mg (Experimental): Participant received 0.0015 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 0.0045 mg (Experimental): Participant received 0.0045 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 0.014 mg (Experimental): Participant received 0.014 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 0.04 mg (Experimental): Participant received 0.04 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 0.12 mg (Experimental): Participant received 0.12 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 0.37 mg (Experimental): Participant received 0.37 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 1.1 mg (Experimental): Participant received 1.1 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 3.3 mg (Experimental): Participant received 3.3 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 10 mg (Experimental): Participant received 10 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 30 mg (Experimental): Participants received 30 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 42 mg (Experimental): Participants received 42 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 59 mg (Experimental): Participants received 59 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 82 mg (Experimental): Participants received 82 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 120 mg (Experimental): Participants received 120 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 170 mg (Experimental): Participants received 170 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 240 mg (Experimental): Participants received 240 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 340 mg (Experimental): Participants received 340 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 480 mg (Experimental): Participants received 480 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 670 mg (Experimental): Participants received 670 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 900 mg (Experimental): Participants received 900 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
  Interventions: Biological: MK-4166
- MK-4166 1.1 mg + Pembro (Experimental): Participants received 1.1 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab
- MK-4166 3.3 mg + Pembro (Experimental): Participants received 3.3 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab
- MK-4166 10 mg + Pembro (Experimental): Participants received 10 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab
- MK-4166 30 mg + Pembro (Experimental): Participants received 30 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab
- MK-4166 42 mg + Pembro (Experimental): Participants received 42 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab
- MK-4166 59 mg + Pembro (Experimental): Participants received 59 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab
- MK-4166 82 mg + Pembro (Experimental): Participants received 82 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab
- MK-4166 120 mg + Pembro (Experimental): Participants received 120 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab
- MK-4166 170 mg + Pembro (Experimental): Participants received 170 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab
- MK-4166 240 mg + Pembro (Experimental): Participants received 240 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab
- MK-4166 340 mg + Pembro (Experimental): Participants received 340 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab
- MK-4166 480 mg + Pembro (Experimental): Participants received 480 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab
- MK-4166 670 mg + Pembro (Experimental): Participants received 670 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab
- MK-4166 900 mg + Pembro (Experimental): Participants received 900 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
  Interventions: Biological: MK-4166; Biological: Pembrolizumab

INTERVENTIONS:
Biological: MK-4166
Biological: Pembrolizumab
  Arms: MK-4166 1.1 mg + Pembro; MK-4166 10 mg + Pembro; MK-4166 120 mg + Pembro; MK-4166 170 mg + Pembro; MK-4166 240 mg + Pembro; MK-4166 3.3 mg + Pembro; MK-4166 30 mg + Pembro; MK-4166 340 mg + Pembro; MK-4166 42 mg + Pembro; MK-4166 480 mg + Pembro; MK-4166 59 mg + Pembro; MK-4166 670 mg + Pembro; MK-4166 82 mg + Pembro; MK-4166 900 mg + Pembro

SUMMARY:
This is planned to be a 5-part dose-escalation study to determine the safety and tolerability of MK-4166 monotherapy and MK-4166 plus pembrolizumab combination therapy, and to establish the maximum tolerated dose (MTD) or maximum administered dose (MAD) of MK-4166 and MK-4166 plus pembrolizumab by defining dose-limiting toxicities (DLTs) in participants with advanced solid tumors.

DETAILED DESCRIPTION:
In Part A, MK-4166 doses will be escalated quickly in successive cohorts and based on safety events may progress to Part B, in which the preliminary MTD will be identified. Based on safety events the study may progress to Part C in which the MTD will be confirmed. In Part D, participants will receive escalating doses of MK-4166 plus a fixed dose of pembrolizumab (MK-3475) 200 mg to determine the MTD for MK-4166 in combination with pembrolizumab. Based on safety events in Part D, the study may progress to Part E in which the MTD for MK-4166 in combination with pembrolizumab will be confirmed.

With Amendments 05/06, the dose confirmation Part C will be removed and the dose confirmation Part E (combination of MK-4166 and pembrolizumab) will be limited to participants with advanced malignant melanoma.

ELIGIBILITY:
Inclusion criteria:

* Has a histologically- or cytologically-confirmed metastatic solid tumor for which there is no available therapy which may convey clinical benefit. Part E: Has advanced malignant melanoma.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Adequate organ function
* Female participants of childbearing potential must have a negative urine or serum pregnancy test and must be surgically sterile or willing to use 2 methods of birth control or abstain from heterosexual activity for the course of the study through 120 days after last dose of study drug
* Male participants must agree to use an adequate method of contraception during sexual contact with females of childbearing potential starting with the first dose of study drug through 180 days after the last dose of study drug
* Submit an evaluable tumor sample for analysis.

Exclusion criteria:

* Chemotherapy, radiation, or biological cancer therapy within 4 weeks prior to the first dose of study drug, or who has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from the adverse events due to cancer therapeutics administered more than 4 weeks earlier
* Currently participating or has participated in a study of an investigational agent or using an investigational device within 28 days of administration of MK-4166
* Expected to require any other form of antineoplastic therapy while on study
* On chronic systemic steroid therapy in excess of replacement doses, or on any other form of immunosuppressive medication
* History of a malignancy for which potentially curative treatment has been completed, with no evidence of malignancy for 5 years excepting successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, or in situ cervical cancer
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Severe hypersensitivity reaction to treatment with another monoclonal antibody
* Active autoimmune disease or a documented history of autoimmune disease, except vitiligo or resolved childhood asthma/atopy
* Active infection requiring therapy
* Current pneumonitis, or a history of (non-infectious) pneumonitis that required steroids
* Prior stem cell or bone marrow transplant
* Positive for human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Regular user (including "recreational use") of any illicit drugs or recent history (within the last year) of substance abuse (including alcohol)
* Symptomatic ascites or pleural effusion
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study
* Clinically significant heart disease
* Major surgery in the past 16 weeks
* Received a live vaccine within 30 days prior to first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Papadopoulos KP, Autio K, Golan T, Dobrenkov K, Chartash E, Chen Q, Wnek R, Long GV. Phase I Study of MK-4166, an Anti-human Glucocorticoid-Induced TNF Receptor Antibody, Alone or with Pembrolizumab in Advanced Solid Tumors. Clin Cancer Res. 2021 Apr 1;27(7):1904-1911. doi: 10.1158/1078-0432.CCR-20-2886. Epub 2020 Dec 21. PMID 33355238

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 116 participants that were non-randomly allocated to treatment, 113 participants received treatment and were evaluable for all analyses.
Period: Overall Study
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 4 | 3 | 3 | 5 | 4 | 3 | 3 | 4 | 3 | 5 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Treated | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 4 | 3 | 3 | 5 | 4 | 3 | 3 | 4 | 3 | 5 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Excluded Medication | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Not completed — Progressive Disease | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 2 | 2 | 3 | 2 | 1 | 2 | 1 | 3 | 1 | 1 | 3 | 2 | 3 | 0 | 1 | 2 | 1 | 2 | 3 | 1 | 1 | 3 | 6
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Transferred to Extension Study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 4 | 3 | 3 | 5 | 4 | 3 | 3 | 4 | 3 | 5 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23 | 116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.0 (0) | 50.0 (0) | 43.0 (0) | 47.0 (0) | 74.0 (0) | 65.0 (0) | 72.0 (0) | 73.0 (0) | 50.0 (0) | 64.7 (9.3) | 57.3 (7.1) | 54.3 (12.6) | 66.8 (22.5) | 61.7 (4.2) | 62.0 (11.8) | 64.6 (11.7) | 66.0 (9.7) | 66.7 (12.1) | 64.0 (12.2) | 71.8 (9.3) | 60.3 (7.0) | 52.2 (17.2) | 58.0 (11.4) | 48.3 (25.5) | 52.3 (3.8) | 74.0 (6.2) | 49.0 (23.2) | 56.3 (11.2) | 63.0 (9.8) | 49.7 (25.1) | 52.7 (17.6) | 63.3 (24.7) | 60.5 (20.5) | 62.0 (15.6) | 60.4 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 3 | 1 | 3 | 3 | 1 | 2 | 1 | 2 | 2 | 1 | 3 | 2 | 1 | 2 | 2 | 2 | 2 | 3 | 3 | 2 | 2 | 1 | 2 | 1 | 6 | 58
  Male | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 1 | 2 | 1 | 4 | 2 | 1 | 2 | 1 | 1 | 4 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 3 | 17 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — 0 participants are reported due to the risk of identification of a person.
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 4 | 3 | 3 | 5 | 4 | 3 | 3 | 4 | 3 | 5 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23 | 116
Race (NIH/OMB) [Count of Participants; unit: Participants] — 0 participants are reported due to the risk of identification of a person.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 4 | 3 | 3 | 5 | 4 | 3 | 3 | 4 | 3 | 5 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23 | 116

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-Limiting Toxicities (DLTs)
Description: DLT's were assessed during the first cycle (21 days) for each dose level and included the following if assessed by the Investigator to be possibly, probably or definitely related to MK-4166 or MK-4166 plus pembrolizumab combination: Grade 4 non-hematologic toxicity; Grade 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia (Grade 4 thrombocytopenia of any duration or Grade 3 thrombocytopenia if associated with bleeding); Grade 3 non-hematologic toxicity lasting >3 days despite optimal supportive care; Grade 3 nausea, vomiting or diarrhea if >3 days despite optimal supportive care; any Grade 3 or Grade 4 non-hematologic laboratory abnormality if medical intervention is required or if leading to hospitalization or if persisting for >1 week; febrile neutropenia Grade 3 or Grade 4; any drug-related AE which caused participant to discontinue treatment during Cycle 1; Grade 5 toxicity; any treatment-related toxicity which caused a >2 week delay in initiation of Cycle 2.
Time Frame: Cycle 1 (up to 21 days)
Population: All allocated participants who received at least 1 dose of study treatment and were evaluable for DLTs in Cycle 1.
Measure: Number; unit: Participants
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE.
  Per protocol, the number of participants experiencing an AE was assessed and reported by arm (MK-4166 monotherapy and MK-4166 plus pembrolizumab combination therapy) as well as by dose cohort.
Time Frame: From first dose up to 90 days post last dose (up to 27 months)
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- MK-4166 Monotherapy: Participants received assigned dose of MK-4166 IV on Day 1 of each 21-day cycle, for up to 4 cycles.
- MK-4166 + Pembro Combination Therapy: Participants received assigned dose of MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles.
Arm/Group | MK-4166 Monotherapy | MK-4166 + Pembro Combination Therapy | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 48 | 65 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Participants | 44 | 63 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 5 | 3 | 3 | 2 | 2 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 22

3. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to AEs
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE.
  Per protocol, the number of participants discontinuing study treatment due to AEs was assessed and reported by arm (MK-4166 monotherapy and MK-4166 plus pembrolizumab combination therapy) as well as by dose cohort.
Time Frame: Up to approximately 24 months
Population: All allocated participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-4166 Monotherapy | MK-4166 + Pembro Combination Therapy | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 48 | 65 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Participants | 2 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 4

4. Secondary Outcome: Maximum Concentration (Cmax) of MK-4166 Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 and plasma isolated for analysis of MK-4166 Cmax. Cmax was defined as the maximum concentration of MK-4166 reached. MK-4166 Cmax was reported by dose cohort. Per protocol, percent geometric coefficient of variation (%GCV) values were not reported for cohorts with n<2 participants.
Time Frame: Cycles 1-4: Day 1 pre-dose, at end of MK-4166 infusion (up to 10 minutes), 2 hours; Days 2, 3, 5 (Cohorts 1-9 only), 8, 15. Each cycle was 21 days. (Up to ~3 months)
Population: All allocated participants who received at least 1 dose of MK-4166 and had evaluable Cmax samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
ng/mL
  Cycle 1 | 0.536 (NA) — NA = %GCV values were not reported when n<2. | 5.18 (NA) — NA = %GCV values were not reported when n<2. | 17.3 (NA) — NA = %GCV values were not reported when n<2. | 21.1 (NA) — NA = %GCV values were not reported when n<2. | 34.3 (NA) — NA = %GCV values were not reported when n<2. | 205 (NA) — NA = %GCV values were not reported when n<2. | 585 (NA) — NA = %GCV values were not reported when n<2. | 1580 (NA) — NA = %GCV values were not reported when n<2. | 3550 (NA) — NA = %GCV values were not reported when n<2. | 10900 (37.1) | 12300 (21.8) | 21800 (13.3) | 23300 (40.7) | 38100 (28.5) | 58600 (16.2) | 68600 (25.1) | 96500 (25.8) | 149000 (16.6) | 195000 (44.4) | 301000 (18.8) | 1790 (16.6) | 3670 (72.9) | 5010 (39.7) | 16300 (32.2) | 16900 (51.1) | 20400 (5.75) | 26300 (32.1) | 28300 (44.5) | 55200 (17.2) | 85900 (12.7) | 109000 (8.9) | 144000 (2.8) | 210000 (11.8) | 234000 (22.7)
  Cycle 2: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 4 | 3 | 2 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 23
  Cycle 2 | 0.0225 (NA) — NA = %GCV values were not reported when n<2. |  |  | 48.2 (NA) — NA = %GCV values were not reported when n<2. | 50.2 (NA) — NA = %GCV values were not reported when n<2. | 533 (NA) — NA = %GCV values were not reported when n<2. |  | 1490 (NA) — NA = %GCV values were not reported when n<2. | 607 (NA) — NA = %GCV values were not reported when n<2. | 11400 (42.0) | 13700 (46.6) | 14400 (92.7) | 31900 (27.2) | 77100 (140.5) | 51500 (38.3) | 115000 (59.1) | 120000 (59.2) | 168000 (20.0) | 228000 (45.7) | 364000 (33.5) | 660 (46.3) | 4010 (11.4) | 541 (31149.1) | 18500 (17.5) | 17900 (52.5) | 27900 (7.4) | 32500 (36.2) | 38100 (25.6) | 65000 (20.7) | 105000 (21.6) | 118000 (14.7) | 175000 (3.2) | 271000 (8.1) | 231000 (173.3)
  Cycle 3: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 3 | 2 | 3 | 3 | 3 | 2 | 3 | 1 | 1 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 18
  Cycle 3 | 0.767 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | 68.8 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | 179 (NA) — NA = %GCV values were not reported when n<2. | 8940 (100.6) | 13400 (37.5) | 16200 (68.9) | 29100 (53.5) | 42000 (16.3) | 52700 (45.8) | 88700 (11.8) | 115000 (49.4) | 147000 (NA) — NA = %GCV values were not reported when n<2. | 247000 (NA) — NA = %GCV values were not reported when n<2. | 389000 (24.4) | 803 (26.2) | 3600 (361.8) | 2190 (263.1) | 18800 (41.8) | 17400 (72.1) | 30300 (11.0) | 37300 (23.4) | 48800 (45.6) | 96800 (62.8) | 111000 (20.6) | 117000 (35.7) | 193000 (18.1) | 321000 (19.3) | 333000 (22.4)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 2 | 0 | 3 | 1 | 2 | 1 | 0 | 2 | 18
  Cycle 4 |  |  |  |  |  |  |  |  |  |  | 7870 (126.1) | 13100 (115.8) | 20800 (44.2) | 38800 (39.1) | 67300 (47.9) | 88800 (18.3) | 86800 (28.8) |  | 256000 (NA) — NA = %GCV values were not reported when n<2. | 501000 (NA) — NA = %GCV values were not reported when n<2. | 42.9 (NA) — NA = %GCV values were not reported when n<2. |  | 10400 (NA) — NA = %GCV values were not reported when n<2. | 14200 (48.0) | 16900 (110.1) | 26600 (12.3) |  | 40600 (43.7) | 43200 (NA) — NA = %GCV values were not reported when n<2. | 126000 (42.5) | 207000 (NA) — NA = %GCV values were not reported when n<2. |  | 318000 (2.0) | 386000 (22.0)

5. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-4166 Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 and plasma isolated for analysis of MK-4166 Tmax. Tmax was defined as time to the maximum concentration of MK-4166 reached. MK-4166 Tmax was reported by dose cohort.
Time Frame: as for outcome 4
Population: All allocated participants who received at least 1 dose of MK-4166 and had evaluable Tmax samples. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Days
  Cycle 1 | 0.96 [0.96 to 0.96] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.03] | 0.08 [0.08 to 0.08] | 0.02 [0.02 to 0.02] | 0.08 [0.08 to 0.08] | 0.05 [0.02 to 0.08] | 0.03 [0.02 to 0.08] | 0.02 [0.02 to 0.03] | 0.02 [0.02 to 0.03] | 0.03 [0.02 to 0.07] | 0.03 [0.02 to 0.03] | 0.03 [0.02 to 1.10] | 0.02 [0.02 to 1.11] | 0.03 [0.02 to 0.08] | 0.02 [0.02 to 0.08] | 0.08 [0.02 to 1.06] | 0.03 [0.03 to 0.08] | 0.03 [0.03 to 0.08] | 0.08 [0.03 to 0.09] | 0.08 [0.03 to 0.09] | 0.02 [0.02 to 0.08] | 0.03 [0.02 to 0.08] | 0.04 [0.02 to 0.08] | 0.03 [0.02 to 0.09] | 0.08 [0.02 to 0.08] | 0.04 [0.03 to 0.08] | 0.03 [0.02 to 0.09] | 0.08 [0.02 to 0.09] | 0.05 [0.02 to 0.13] | 0.08 [0.02 to 0.13]
  Cycle 2: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 4 | 3 | 2 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 23
  Cycle 2 | 6.98 [6.98 to 6.98] |  |  | 0.03 [0.03 to 0.03] | 0.04 [0.04 to 0.04] | 0.02 [0.02 to 0.02] |  | 0.02 [0.02 to 0.02] | 0.03 [0.03 to 0.03] | 0.03 [0.02 to 0.08] | 0.03 [0.03 to 0.08] | 0.05 [0.02 to 0.08] | 0.03 [0.02 to 0.08] | 0.02 [0.02 to 0.03] | 0.07 [0.02 to 0.08] | 0.47 [0.02 to 0.91] | 0.02 [0.02 to 0.09] | 0.03 [0.02 to 0.08] | 0.02 [0.02 to 0.08] | 0.02 [0.02 to 0.08] | 0.03 [0.02 to 0.08] | 0.03 [0.03 to 0.03] | 0.02 [0.02 to 0.1] | 0.02 [0.02 to 0.9] | 0.08 [0.02 to 0.08] | 0.05 [0.02 to 0.08] | 0.03 [0.02 to 0.03] | 0.02 [0.02 to 0.08] | 0.03 [0.02 to 0.90] | 0.08 [0.03 to 0.08] | 0.02 [0.02 to 0.08] | 0.08 [0.08 to 0.08] | 0.06 [0.03 to 0.08] | 0.08 [0.02 to 1.08]
  Cycle 3: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 3 | 2 | 3 | 3 | 3 | 2 | 3 | 1 | 1 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 18
  Cycle 3 | 0.08 [0.08 to 0.08] |  |  |  | 0.04 [0.04 to 0.04] |  |  |  | 0.03 [0.03 to 0.03] | 0.03 [0.02 to 0.08] | 0.02 [0.02 to 0.08] | 0.05 [0.02 to 0.08] | 0.03 [0.02 to 0.09] | 0.02 [0.02 to 0.08] | 0.02 [0.02 to 0.07] | 0.08 [0.08 to 0.08] | 0.08 [0.02 to 0.08] | 0.08 [0.08 to 0.08] | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.08] | 0.03 [0.03 to 0.03] | 0.03 [0.03 to 0.03] | 0.06 [0.04 to 0.09] | 0.02 [0.02 to 0.11] | 0.08 [0.02 to 0.08] | 0.03 [0.02 to 0.03] | 0.08 [0.03 to 0.08] | 0.03 [0.02 to 0.08] | 0.08 [0.02 to 0.08] | 0.02 [0.02 to 0.08] | 0.02 [0.02 to 0.09] | 0.05 [0.02 to 0.08] | 0.02 [0.02 to 0.02] | 0.03 [0.02 to 0.09]
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 2 | 0 | 3 | 1 | 2 | 1 | 0 | 2 | 18
  Cycle 4 |  |  |  |  |  |  |  |  |  |  | 0.06 [0.03 to 0.08] | 0.03 [0.02 to 0.03] | 0.02 [0.02 to 0.02] | 0.05 [0.02 to 0.08] | 0.02 [0.02 to 0.02] | 0.03 [0.02 to 0.03] | 0.06 [0.02 to 0.09] |  | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.02] | 0.03 [0.03 to 0.03] |  | 0.09 [0.09 to 0.09] | 0.08 [0.08 to 0.08] | 0.05 [0.02 to 0.08] | 0.02 [0.02 to 0.03] |  | 0.08 [0.03 to 0.08] | 0.02 [0.02 to 0.02] | 0.05 [0.02 to 0.09] | 0.02 [0.02 to 0.02] |  | 0.08 [0.08 to 0.08] | 0.08 [0.02 to 0.09]

6. Secondary Outcome: Terminal Half-Life (t ½) of MK-4166 Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 and plasma isolated for analysis of MK-4166 t½. t½ was defined as the time required to divide the MK-4166 plasma concentration by two after reaching pseudo-equilibrium, following a single dose of MK-4166. MK-4166 t½ was reported by dose cohort. Per protocol, % GCV values were not reported for cohorts with n<2 participants.
Time Frame: as for outcome 4
Population: All allocated participants who received at least 1 dose of MK-4166 and had evaluable t½ samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Days
  Cycle 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 4 | 23
  Cycle 1 | 2.61 (NA) — NA = %GCV values were not reported when n<2. | 2.74 (NA) — NA = %GCV values were not reported when n<2. | 2.68 (NA) — NA = %GCV values were not reported when n<2. | 3.48 (NA) — NA = %GCV values were not reported when n<2. | 2.73 (NA) — NA = %GCV values were not reported when n<2. | 2.10 (NA) — NA = %GCV values were not reported when n<2. | 3.39 (NA) — NA = %GCV values were not reported when n<2. | 3.30 (NA) — NA = %GCV values were not reported when n<2. | 7.62 (NA) — NA = %GCV values were not reported when n<2. | 7.7 (67.2) | 7.49 (107.2) | 2.93 (85.2) | 12.8 (27.6) | 6.37 (87.7) | 7.66 (31.4) | 5.17 (126.5) | 12.0 (69.2) | 11.3 (22.7) | 13.1 (37.2) | 12.3 (4.5) | 2.86 (9.63) | 3.64 (27.7) | 6.15 (78.5) | 12.0 (60.9) | 7.31 (48.9) | 8.60 (66.6) | 8.84 (14.3) | 10.9 (28.8) | 11.9 (12.0) | 13.0 (10.6) | 7.81 (120.0) | 13.4 (37.4) | 9.03 (77.4) | 12.0 (70.1)
  Cycle 2: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 4 | 3 | 2 | 3 | 3 | 2 | 2 | 3 | 2 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 20
  Cycle 2 | NA (NA) — NA = t½ was not calculable. |  |  | 2.31 (NA) — NA = %GCV values were not reported when n<2. | 3.22 (NA) — NA = %GCV values were not reported when n<2. | 3.42 (NA) — NA = %GCV values were not reported when n<2. |  | 1.88 (NA) — NA = %GCV values were not reported when n<2. | NA (NA) — NA = t½ was not calculable. | 4.53 (171.6) | 7.21 (167.8) | 1.31 (2100.9) | 9.95 (38.4) | 5.82 (65.6) | 8.97 (39.5) | 11.4 (123.7) | 13.1 (32.8) | 10.2 (13.0) | 11.2 (49.6) | 14.1 (36.7) | 3.74 (486.6) | 1.38 (158.1) | 4.55 (318) | 10.5 (62.9) | 6.92 (82.0) | 5.82 (33.3) | 11.7 (14.3) | 9.22 (106.0) | 12.4 (36.6) | 15.7 (10.9) | 7.43 (111.8) | 11.7 (12.3) | 16.2 (5.36) | 13.2 (56.4)
  Cycle 3: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 3 | 3 | 3 | 2 | 3 | 1 | 1 | 2 | 3 | 2 | 1 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 1 | 2 | 18
  Cycle 3 | 3.34 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | 1.76 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | NA (NA) — NA = t½ was not calculable. | 3.11 (120.5) | 4.52 (376.5) | 11.9 (NA) — NA = %GCV values were not reported when n<2. | 6.54 (54.0) | 9.59 (44.8) | 3.61 (787.8) | 11.9 (12.4) | 11.9 (29.2) | 11.3 (NA) — NA = %GCV values were not reported when n<2. | 10.4 (NA) — NA = %GCV values were not reported when n<2. | 21.4 (60) | 2.19 (394.0) | 3.72 (88.5) | 16.6 (NA) — NA = %GCV values were not reported when n<2. | 10.4 (95.0) | 7.32 (92.3) | 5.10 (23.4) | 7.91 (23.9) | 9.97 (30.5) | 12.3 (46.1) | 22.1 (50.8) | 5.75 (269.1) | 17.6 (NA) — NA = %GCV values were not reported when n<2. | 15.7 (18.6) | 21.6 (85.4)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 2 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 3 | 1 | 2 | 1 | 0 | 1 | 16
  Cycle 4 |  |  |  |  |  |  |  |  |  |  | 2.04 (706.9) | 8.79 (NA) — NA = %GCV values were not reported when n<2. | 2.59 (220.3) | NA (NA) — NA = t½ was not calculable. | 7.43 (139.3) | 8.14 (11.5) | 17.8 (NA) — NA = %GCV values were not reported when n<2. |  | 3.91 (NA) — NA = %GCV values were not reported when n<2. | NA — NA = %GCV values were not reported when n<2. | NA — NA = t½ was not calculable. |  | 7.12 (NA) — NA = %GCV values were not reported when n<2. | 6.68 (103.1) | 13.1 (NA) — NA = %GCV values were not reported when n<2. | 6.27 (8.1) |  | 13.8 (34.5) | 14.8 (NA) — NA = %GCV values were not reported when n<2. | 16.4 (27.6) | 13.0 (NA) — NA = %GCV values were not reported when n<2. |  | 12.0 (NA) — NA = %GCV values were not reported when n<2. | 17.2 (48.6)

7. Secondary Outcome: Area Under the Concentration-Time Curve of MK-4166 From Time Zero to 21 Hours After Dosing (AUC 0-21) Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 and plasma isolated for analysis of MK-4166 AUC0-21. AUC0-21 was defined as the area under the concentration-time curve of MK-4166 from time zero to 21 hours after dosing. MK-4166 AUC0-21 was reported by dose cohort. Per protocol, % GCV values were not reported for cohorts with n<2 participants.
Time Frame: Cycles 1-4: Day 1 pre-dose, at end of MK-4166 infusion (up to 10 minutes), 2 hours; Day 2. Each cycle was 21 days. (Up to ~3 months)
Population: All allocated participants who received at least 1 dose of MK-4166 and had evaluable AUC0-21 samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days•ng/mL
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Days•ng/mL
  Cycle 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 4 | 23
  Cycle 1 | 1.08 (NA) — NA = %GCV values were not reported when n<2. | 3.91 (NA) — NA = %GCV values were not reported when n<2. | 24.7 (NA) — NA = %GCV values were not reported when n<2. | 39.0 (NA) — NA = %GCV values were not reported when n<2. | 69.4 (NA) — NA = %GCV values were not reported when n<2. | 672 (NA) — NA = %GCV values were not reported when n<2. | 3140 (NA) — NA = %GCV values were not reported when n<2. | 8300 (NA) — NA = %GCV values were not reported when n<2. | 19100 (NA) — NA = %GCV values were not reported when n<2. | 84700 (36.5) | 111000 (32.9) | 142000 (31.1) | 226000 (46.3) | 291000 (39.6) | 457000 (23.3) | 426000 (30.4) | 770000 (59.0) | 1110000 (21.4) | 1730000 (28.7) | 3110000 (17.5) | 7700 (32.6) | 19900 (87.1) | 33800 (89.1) | 137000 (41.4) | 119000 (71.4) | 147000 (25.9) | 271000 (25) | 248000 (57.6) | 516000 (21.1) | 832000 (11.4) | 986000 (26.2) | 137000 (7.7) | 1740000 (50.3) | 2130000 (27.5)
  Cycle 2: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 4 | 3 | 2 | 3 | 3 | 2 | 2 | 3 | 2 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 20
  Cycle 2 | 0.141 (NA) — NA = %GCV values were not reported when n<2. |  |  | 126 (NA) — NA = %GCV values were not reported when n<2. | 118 (NA) — NA = %GCV values were not reported when n<2. | 2610 (NA) — NA = %GCV values were not reported when n<2. |  | 3510 (NA) — NA = %GCV values were not reported when n<2. | NA (NA) — NA = %GCV values were not reported when n<2. | 48600 (226.2) | 51800 (660.7) | 14500 (19927.0) | 273000 (50.1) | 223000 (45.6) | 401000 (55.9) | 860000 (53.4) | 1160000 (72.1) | 1590000 (33.3) | 2090000 (19.8) | 4580000 (21.1) | 1120 (120.6) | 7330 (150.8) | 6380 (503154.6) | 167000 (56.9) | 116000 (121.4) | 216000 (32.4) | 278000 (37.1) | 279000 (84.3) | 594000 (27.1) | 1170000 (15.1) | 678000 (305.7) | 1760000 (11.9) | 3280000 (5.08) | 2880000 (49.0)
  Cycle 3: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 3 | 3 | 3 | 2 | 3 | 1 | 1 | 2 | 3 | 2 | 1 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 1 | 2 | 18
  Cycle 3 | 0.893 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | 135 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | NA (NA) — NA = AUC0-21 was not calculable. | 17400 (711.2) | 55700 (733.9) | 235000 (NA) — NA = %GCV values were not reported when n<2. | 217000 (87.0) | 306000 (32.2) | 173000 (658.5) | 749000 (6.8) | 1180000 (69.4) | 1370000 (NA) — NA = %GCV values were not reported when n<2. | 2390000 (NA) — NA = %GCV values were not reported when n<2. | 5410000 (4.01) | 1110 (104.1) | 33900 (8.86) | 79300 (NA) — NA = %GCV values were not reported when n<2. | 182000 (81.4) | 123000 (156.1) | 152000 (11.5) | 301000 (27.7) | 330000 (79.3) | 631000 (10.4) | 1310000 (18.8) | 692000 (277.7) | 2220000 (NA) — NA = %GCV values were not reported when n<2. | 3440000 (7.9) | 3790000 (28.7)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 2 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 3 | 1 | 2 | 1 | 0 | 1 | 16
  Cycle 4 |  |  |  |  |  |  |  |  |  |  | 18500 (8160.0) | 250000 (NA) — NA = %GCV values were not reported when n<2. | 80600 (247.9) | NA (NA) — NA = AUC0-21 was not calculable. | 503000 (133.9) | 716000 (0.359) | 1410000 (NA) — NA = %GCV values were not reported when n<2. |  | 1400000 (NA) — NA = %GCV values were not reported when n<2. | NA — NA = AUC0-21 was not calculable. | NA — NA = AUC0-21 was not calculable. |  | 80400 (NA) — NA = %GCV values were not reported when n<2. | 107000 (136.8) | 353000 (NA) — NA = %GCV values were not reported when n<2. | 148000 (24.9) |  | 394000 (66.0) | 575000 (NA) — NA = %GCV values were not reported when n<2. | 1580000 (46.2) | 2350000 (NA) — NA = %GCV values were not reported when n<2. |  | 3800000 (NA) — NA = %GCV values were not reported when n<2. | 4360000 (33.7)

8. Secondary Outcome: Area Under the Concentration-Time Curve of MK-4166 From Time Zero to The Last Quantifiable Sample (AUC 0-last) Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 and plasma isolated for analysis of MK-4166 AUC0-last. AUC0-last was defined as the area under the concentration-time curve of MK-4166 from time zero to the last quantifiable sample. MK-4166 AUC0-last was reported by dose cohort. Per protocol, % GCV values were not reported for cohorts with n<2 participants.
Time Frame: as for outcome 4
Population: All allocated participants who received at least 1 dose of MK-4166 and had evaluable AUC0-last samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days•ng/mL
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Days•ng/mL
  Cycle 1 | 1.08 (NA) — NA = %GCV values were not reported when n<2. | 3.89 (NA) — NA = %GCV values were not reported when n<2. | 24.6 (NA) — NA = %GCV values were not reported when n<2. | 39.0 (NA) — NA = %GCV values were not reported when n<2. | 69.4 (NA) — NA = %GCV values were not reported when n<2. | 672 (NA) — NA = %GCV values were not reported when n<2. | 3010 (NA) — NA = %GCV values were not reported when n<2. | 8300 (NA) — NA = %GCV values were not reported when n<2. | 14300 (NA) — NA = %GCV values were not reported when n<2. | 79500 (34.6) | 111000 (32.7) | 141000 (31.6) | 226000 (46.4) | 290000 (39.4) | 451000 (23.9) | 354000 (51.6) | 677000 (82.2) | 1170000 (31.1) | 1720000 (29.0) | 3310000 (17.1) | 7700 (32.6) | 14100 (57.6) | 31900 (88.8) | 137000 (41.5) | 120000 (71.0) | 142000 (31.9) | 200000 (76.6) | 248000 (57.5) | 477000 (16.2) | 830000 (11.3) | 967000 (25.3) | 738000 (141.5) | 1280000 (126.2) | 2140000 (27.5)
  Cycle 2: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 4 | 3 | 2 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 23
  Cycle 2 | 0.0632 (NA) — NA = %GCV values were not reported when n<2. |  |  | 86.9 (NA) — NA = %GCV values were not reported when n<2. | 118 (NA) — NA = %GCV values were not reported when n<2. | 2010 (NA) — NA = %GCV values were not reported when n<2. |  | 1780 (NA) — NA = %GCV values were not reported when n<2. | 21.1 (NA) — NA = %GCV values were not reported when n<2. | 48600 (226.2) | 51600 (660.6) | 14400 (20883.7) | 268000 (49.1) | 223000 (45.3) | 128000 (759.0) | 864000 (54.7) | 1160000 (72.3) | 635000 (247.7) | 1790000 (31.7) | 2620000 (116.6) | 1110 (118.9) | 6510 (182.3) | 309 (4954684876.5) | 167000 (56.9) | 115000 (121.4) | 228000 (40.9) | 280000 (35.7) | 280000 (83.6) | 616000 (25.9) | 1170000 (13.7) | 681000 (307.0) | 1710000 (15.7) | 3770000 (25.4) | 1710000 (371.9)
  Cycle 3: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 3 | 2 | 3 | 3 | 3 | 2 | 3 | 1 | 1 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 18
  Cycle 3 | 0.879 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | 135 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | 7.48 (NA) — NA = %GCV values were not reported when n<2. | 19600 (351.9) | 51400 (640.7) | 25300 (14504.2) | 172000 (69.1) | 281000 (19.5) | 168000 (728.3) | 756000 (5.0) | 1110000 (59.1) | 1110000 (NA) — NA = %GCV values were not reported when n<2. | 2400000 (NA) — NA = %GCV values were not reported when n<2. | 1910000 (294) | 740 (53.9) | 4070 (18558.6) | 5130 (177486.3) | 162000 (63.3) | 118000 (153.4) | 153000 (12.2) | 219000 (18.5) | 323000 (80.9) | 579000 (14.8) | 638000 (195.6) | 443000 (353.2) | 473000 (480.0) | 3480000 (6.2) | 3920000 (29.1)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 2 | 0 | 3 | 1 | 2 | 1 | 0 | 2 | 18
  Cycle 4 |  |  |  |  |  |  |  |  |  |  | 11500 (4140.6) | 14600 (18895.8) | 61500 (136.5) | 79100 (265.0) | 184000 (174.6) | 379000 (5.5) | 254000 (175.0) |  | 433000 (NA) — NA = %GCV values were not reported when n<2. | 469000 (NA) — NA = %GCV values were not reported when n<2. | 1.72 (NA) — NA = %GCV values were not reported when n<2. |  | 46000 (NA) — NA = %GCV values were not reported when n<2. | 80800 (140.8) | 12600 (1377431.1) | 142000 (39.4) |  | 365000 (44.1) | 574000 (NA) — NA = %GCV values were not reported when n<2. | 1580000 (46.6) | 2280000 (NA) — NA = %GCV values were not reported when n<2. |  | 975000 (99.2) | 2750000 (135.4)

9. Secondary Outcome: Area Under the Concentration-Time Curve of MK-4166 From Time Zero to Infinity (AUC 0-inf) Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 and plasma isolated for analysis of MK-4166 AUC0-inf. AUC0-inf was defined as the area under the concentration-time curve of MK-4166 from time zero to infinity. MK-4166 AUC0-inf was reported by dose cohort. Per protocol, % GCV values were not reported for cohorts with n<2 participants.
Time Frame: as for outcome 4
Population: All allocated participants who received at least 1 dose of MK-4166 and had evaluable AUC0-inf samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days•ng/mL
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Days•ng/mL
  Cycle 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 4 | 23
  Cycle 1 | 1.09 (NA) — NA = %GCV values were not reported when n<2. | 3.92 (NA) — NA = %GCV values were not reported when n<2. | 24.8 (NA) — NA = %GCV values were not reported when n<2. | 39.3 (NA) — NA = %GCV values were not reported when n<2. | 69.5 (NA) — NA = %GCV values were not reported when n<2. | 673 (NA) — NA = %GCV values were not reported when n<2. | 3190 (NA) — NA = %GCV values were not reported when n<2. | 8420 (NA) — NA = %GCV values were not reported when n<2. | 29400 (NA) — NA = %GCV values were not reported when n<2. | 105000 (54) | 141000 (55.5) | 148000 (37.7) | 333000 (59.5) | 345000 (54.4) | 558000 (31.1) | 501000 (51.5) | 1120000 (67.1) | 1500000 (17.2) | 2580000 (9.88) | 4520000 (19.2) | 7750 (32.8) | 20600 (89.4) | 40200 (121.9) | 200000 (74.6) | 142000 (90.1) | 187000 (46.0) | 336000 (23.4) | 338000 (76.2) | 730000 (15.9) | 1240000 (12.4) | 1300000 (52.3) | 2090000 (26.2) | 2340000 (77.0) | 3200000 (43.0)
  Cycle 2: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 4 | 3 | 2 | 3 | 3 | 2 | 2 | 3 | 2 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 20
  Cycle 2 | NA (NA) — NA = AUC0-inf was not calculable. |  |  | 126 (NA) — NA = %GCV values were not reported when n<2. | 118 (NA) — NA = %GCV values were not reported when n<2. | 2660 (NA) — NA = %GCV values were not reported when n<2. |  | 3490 (NA) — NA = %GCV values were not reported when n<2. | NA (NA) — NA = AUC0-inf was not calculable. | 58600 (326.9) | 68800 (1111.6) | 15400 (28630.7) | 360000 (68.6) | 252000 (59.2) | 503000 (78.7) | 1280000 (6.1) | 1740000 (71.9) | 2090000 (39.2) | 2950000 (4.1) | 7270000 (0.2) | 1550 (49.7) | 7010 (176.2) | 7660 (2164569.0) | 232000 (92.0) | 141000 (168.9) | 238000 (40.4) | 392000 (38.9) | 385000 (150.0) | 849000 (15.3) | 1930000 (20.7) | 874000 (450.1) | 2500000 (18.6) | 5570000 (8.3) | 4520000 (70.6)
  Cycle 3: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 3 | 3 | 3 | 2 | 3 | 1 | 1 | 2 | 3 | 2 | 1 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 1 | 2 | 18
  Cycle 3 | 0.896 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | 135 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | NA (NA) — NA = AUC0-inf was not calculable. | 18700 (896.0) | 70000 (1119.8) | 330000 (NA) — NA = %GCV values were not reported when n<2. | 251000 (105.1) | 396000 (53.5) | 216000 (1232.6) | 1050000 (2.7) | 1690000 (69.9) | 1880000 (NA) — NA = %GCV values were not reported when n<2. | 3190000 (NA) — NA = %GCV values were not reported when n<2. | 11300000 (33.8) | 1210 (104.1) | 35700 (1.4) | 136000 (NA) — NA = %GCV values were not reported when n<2. | 261000 (123.7) | 155000 (236.1) | 162000 (15.6) | 360000 (28.9) | 430000 (86.6) | 915000 (17.1) | 2740000 (52.3) | 909000 (438.2) | 3910000 (NA) — NA = %GCV values were not reported when n<2. | 5690000 (2.23) | 8000000 (82.8)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 2 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 3 | 1 | 2 | 1 | 0 | 1 | 16
  Cycle 4 |  |  |  |  |  |  |  |  |  |  | 18200 (20134.8) | 309000 (NA) — NA = %GCV values were not reported when n<2. | 85500 (284.2) | NA (NA) — NA = AUC0-inf was not calculable. | 644000 (228.9) | 862000 (4.6) | 2520000 (NA) — NA = %GCV values were not reported when n<2. |  | 1460000 (NA) — NA = %GCV values were not reported when n<2. | NA (NA) — NA = AUC0-inf was not calculable. | NA (NA) — NA = AUC0-inf was not calculable. |  | 92300 (NA) — NA = %GCV values were not reported when n<2. | 129000 (200.9) | 524000 (NA) — NA = %GCV values were not reported when n<2. | 164000 (22.9) |  | 609000 (96.4) | 914000 (NA) — NA = %GCV values were not reported when n<2. | 2720000 (67.4) | 3480000 (NA) — NA = %GCV values were not reported when n<2. |  | 5400000 (NA) — NA = %GCV values were not reported when n<2. | 7910000 (54.9)

10. Secondary Outcome: Apparent Clearance (CL) of MK-4166 Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 and plasma isolated for analysis of MK-4166 CL. CL was defined as the volume of plasma from which MK-4166 is eliminated per unit time following IV MK-4166 administration. MK-4166 CL was reported by dose cohort. Per protocol, % GCV values were not reported for cohorts with n<2 participants.
Time Frame: as for outcome 4
Population: All allocated participants who received at least 1 dose of MK-4166 and had evaluable CL samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)/day
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Liters (L)/day
  Cycle 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 4 | 23
  Cycle 1 | 1.38 (NA) — NA = %GCV values were not reported when n<2. | 1.15 (NA) — NA = %GCV values were not reported when n<2. | 0.565 (NA) — NA = %GCV values were not reported when n<2. | 1.02 (NA) — NA = %GCV values were not reported when n<2. | 1.73 (NA) — NA = %GCV values were not reported when n<2. | 0.550 (NA) — NA = %GCV values were not reported when n<2. | 0.344 (NA) — NA = %GCV values were not reported when n<2. | 0.392 (NA) — NA = %GCV values were not reported when n<2. | 0.341 (NA) — NA = %GCV values were not reported when n<2. | 0.286 (54.0) | 0.299 (55.5) | 0.400 (37.7) | 0.246 (59.5) | 0.348 (54.4) | 0.305 (31.1) | 0.479 (51.5) | 0.304 (67.1) | 0.320 (17.2) | 0.259 (9.9) | 0.199 (19.2) | 0.142 (32.8) | 0.161 (89.4) | 0.249 (122) | 0.150 (74.4) | 0.296 (90.1) | 0.315 (46.0) | 0.244 (23.4) | 0.302 (51.3) | 0.233 (15.9) | 0.193 (12.4) | 0.262 (52.3) | 0.230 (26.2) | 0.287 (77.0) | 0.279 (40.9)
  Cycle 2: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 4 | 3 | 2 | 3 | 3 | 2 | 2 | 3 | 2 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 20
  Cycle 2 | 10.6 (NA) — NA = %GCV values were not reported when n<2. |  |  | 0.319 (NA) — NA = %GCV values were not reported when n<2. | 1.02 (NA) — NA = %GCV values were not reported when n<2. | 0.142 (NA) — NA = %GCV values were not reported when n<2. |  | 0.940 (NA) — NA = %GCV values were not reported when n<2. | NA (NA) — NA = CL was not calculable. | 0.617 (226.2) | 0.811 (660.7) | 4.06 (19927.0) | 0.301 (50.1) | 0.538 (45.6) | 0.424 (55.9) | 0.279 (53.4) | 0.293 (72.1) | 0.302 (33.3) | 0.321 (19.8) | 0.197 (21.1) | 0.98 (120.6) | 0.450 (150.8) | 1.57 (503154.6) | 0.182 (60.1) | 0.362 (121.4) | 0.273 (32.4) | 0.294 (37.1) | 0.430 (84.3) | 0.286 (27.1) | 0.205 (15.1) | 0.502 (305.7) | 0.272 (11.9) | 0.204 (5.1) | 0.313 (49.0)
  Cycle 3: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 3 | 3 | 3 | 2 | 3 | 1 | 1 | 2 | 3 | 2 | 1 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 1 | 2 | 18
  Cycle 3 | 1.68 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | 0.887 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | NA (NA) — NA = CL was not calculable. | 1.73 (711.2) | 0.754 (733.9) | 0.251 (NA) — NA = %GCV values were not reported when n<2. | 0.378 (87.0) | 0.392 (32.2) | 0.982 (658.5) | 0.321 (6.8) | 0.288 (69.4) | 0.349 (NA) — NA = %GCV values were not reported when n<2. | 0.280 (NA) — NA = %GCV values were not reported when n<2. | 0.166 (4.0) | 0.987 (104.1) | 0.0973 (8.86) | 0.126 (NA) — NA = %GCV values were not reported when n<2. | 0.165 (81.4) | 0.341 (156.1) | 0.388 (11.5) | 0.273 (27.7) | 0.364 (79.3) | 0.269 (10.4) | 0.183 (18.8) | 0.491 (277.7) | 0.217 (NA) — NA = %GCV values were not reported when n<2. | 0.195 (7.9) | 0.238 (28.7)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 2 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 3 | 1 | 2 | 1 | 0 | 1 | 16
  Cycle 4 |  |  |  |  |  |  |  |  |  |  | 2.27 (8160.0) | 0.236 (NA) — NA = %GCV values were not reported when n<2. | 1.02 (247.9) | NA (NA) — NA = CL was not calculable. | 0.338 (133.9) | 0.335 (0.4) | 0.241 (NA) — NA = %GCV values were not reported when n<2. |  | 0.477 (NA) — NA = %GCV values were not reported when n<2. | NA (NA) — NA = CL was not calculable. | NA (NA) — NA = CL was not calculable. |  | 0.124 (NA) — NA = %GCV values were not reported when n<2. | 0.282 (136.8) | 0.119 (NA) — NA = %GCV values were not reported when n<2. | 0.398 (24.9) |  | 0.305 (66.0) | 0.296 (NA) — NA = %GCV values were not reported when n<2. | 0.152 (46.2) | 0.145 (NA) — NA = %GCV values were not reported when n<2. |  | 0.176 (NA) — NA = %GCV values were not reported when n<2. | 0.206 (33.7)

11. Secondary Outcome: Apparent Volume of Distribution (V) of MK-4166 Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 and plasma isolated for analysis of MK-4166 V. V was defined as the theoretical volume that would be necessary to contain the total amount of administered MK-4166 at the same concentration that it is observed in the blood plasma. MK-4166 V was reported by dose cohort. Per protocol, % GCV values were not reported for cohorts with n<2 participants.
Time Frame: as for outcome 4
Population: All allocated participants who received at least 1 dose of MK-4166 and had evaluable V samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Liters
  Cycle 1: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 6 | 3 | 3 | 3 | 3 | 3 | 5 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 4 | 23
  Cycle 1 | 5.19 (NA) — NA = %GCV values were not reported when n<2. | 4.55 (NA) — NA = %GCV values were not reported when n<2. | 2.18 (NA) — NA = %GCV values were not reported when n<2. | 5.11 (NA) — NA = %GCV values were not reported when n<2. | 6.80 (NA) — NA = %GCV values were not reported when n<2. | 1.67 (NA) — NA = %GCV values were not reported when n<2. | 1.68 (NA) — NA = %GCV values were not reported when n<2. | 1.87 (NA) — NA = %GCV values were not reported when n<2. | 3.74 (NA) — NA = %GCV values were not reported when n<2. | 3.20 (32.6) | 3.23 (48.9) | 1.69 (49.7) | 4.56 (35.4) | 3.19 (69.7) | 3.37 (19.3) | 3.57 (79.9) | 5.27 (67.9) | 5.21 (34.4) | 4.92 (48.4) | 3.54 (17.1) | 0.587 (30.2) | 0.844 (55.6) | 2.21 (33.9) | 2.61 (10.8) | 3.12 (46.6) | 3.91 (22.6) | 3.11 (28.8) | 4.73 (21.2) | 4.01 (27.1) | 3.62 (14.0) | 2.95 (48.8) | 4.44 (10.4) | 3.74 (1.0) | 4.85 (38.1)
  Cycle 2: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 4 | 3 | 1 | 3 | 3 | 2 | 2 | 3 | 2 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 20
  Cycle 2 | NA (NA) — NA = V was not calculable. |  |  | 1.10 (NA) — NA = %GCV values were not reported when n<2. | 2.49 (NA) — NA = %GCV values were not reported when n<2. | 0.722 (NA) — NA = %GCV values were not reported when n<2. |  | 2.41 (NA) — NA = %GCV values were not reported when n<2. | NA (NA) — NA = V was not calculable. | 3.75 (27.1) | 6.59 (46.1) | 3.91 (NA) — NA = %GCV values were not reported when n<2. | 4.25 (11.0) | 4.40 (14.9) | 5.10 (2.5) | 4.41 (263.0) | 5.44 (88.1) | 4.42 (21.1) | 5.19 (75.3) | 4.11 (63.3) | 5.61 (3589.3) | 0.870 (13.1) | 2.97 (96.8) | 2.76 (3.1) | 3.67 (35.8) | 2.41 (3.0) | 4.9 (40.3) | 5.89 (18.4) | 4.77 (58.9) | 4.58 (10.6) | 4.36 (23.7) | 4.68 (2.0) | 4.83 (0.5) | 5.94 (36.7)
  Cycle 3: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 3 | 3 | 2 | 2 | 3 | 1 | 1 | 2 | 2 | 2 | 1 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 1 | 2 | 18
  Cycle 3 | 3.58 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | 1.99 (NA) — NA = %GCV values were not reported when n<2. |  |  |  | NA (NA) — NA = V was not calculable. | 6.13 (84.5) | 4.76 (34.1) | 4.15 (NA) — NA = %GCV values were not reported when n<2. | 3.62 (28.9) | 5.14 (17.2) | 5.54 (8.6) | 5.25 (11.9) | 4.87 (83.3) | 5.53 (NA) — NA = %GCV values were not reported when n<2. | 4.24 (NA) — NA = %GCV values were not reported when n<2. | 5.2 (61.6) | 5.45 (862.6) | 0.499 (111.2) | 3.01 (NA) — NA = %GCV values were not reported when n<2. | 2.5 (42.7) | 3.56 (62.3) | 2.90 (8.8) | 3.10 (39.1) | 4.96 (69.5) | 4.62 (50.2) | 5.7 (25.2) | 3.97 (12.2) | 5.41 (NA) — NA = %GCV values were not reported when n<2. | 4.38 (25.2) | 7.23 (61.1)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 3 | 1 | 2 | 1 | 0 | 1 | 16
  Cycle 4 |  |  |  |  |  |  |  |  |  |  | 3.32 (NA) — NA = %GCV values were not reported when n<2. | 3.00 (NA) — NA = %GCV values were not reported when n<2. | 4.03 (16.5) | NA (NA) — NA = V was not calculable. | 3.55 (5.0) | 3.97 (12.0) | 6.16 (NA) — NA = %GCV values were not reported when n<2. |  | 2.82 (NA) — NA = %GCV values were not reported when n<2. | NA (NA) — NA = V was not calculable. | NA (NA) — NA = V was not calculable. |  | 1.27 (NA) — NA = %GCV values were not reported when n<2. | 2.71 (16.6) | 2.22 (NA) — NA = %GCV values were not reported when n<2. | 3.49 (32.9) |  | 5.93 (23.7) | 6.29 (NA) — NA = %GCV values were not reported when n<2. | 3.61 (16.4) | 2.72 (NA) — NA = %GCV values were not reported when n<2. |  | 3.04 (NA) — NA = %GCV values were not reported when n<2. | 5.14 (37.4)

12. Secondary Outcome: Maximum Concentration (Cmax) of Pembrolizumab Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 from MK-4166 plus pembrolizumab combination cohorts only and plasma isolated for analysis of pembrolizumab Cmax. Cmax was defined as the maximum concentration of pembrolizumab reached. Pembrolizumab Cmax was reported by dose cohort for all participants that received MK-4166 plus pembrolizumab combination therapy. Per protocol, participants receiving MK-4166 monotherapy were excluded from this analysis.
Time Frame: Cycles 1-4: Day 1 pre-dose, at end of pembro infusion (up to 10 minutes), at end of MK-4166 infusion (up to 10 minutes), ~2 hours after start of MK-4166 infusion, Days 2, 3, 8, 15. Each cycle was 21 days. (Up to ~3 months)
Population: All allocated participants who received ≥1 dose of pembrolizumab and had evaluable Cmax samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants, and MK-4166 monotherapy dose cohorts were not analyzed. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
ng/mL
  Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 2 | 3 | 3 | 4 | 23
  Cycle 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 82400 (27.9) | 68500 (32.4) | 51700 (25.7) | 81700 (17.2) | 57600 (35.7) | 78400 (18.4) | 72600 (24.3) | 57700 (27.2) | 63300 (30.7) | 83700 (24.8) | 66900 (4.1) | 81600 (22.5) | 70400 (15.1) | 69900 (20.9)
  Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 2 | 3 | 2 | 2 | 23
  Cycle 2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 90000 (32.2) | 76800 (31.8) | 61300 (17.2) | 16200 (109.6) | 73000 (35.9) | 96800 (14.2) | 85700 (40.7) | 48700 (79.3) | 78500 (12.5) | 82300 (25.5) | 86000 (17.4) | 96600 (4.9) | 94100 (12.9) | 80100 (25.4)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 2 | 18
  Cycle 3 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 97200 (56.3) | 78400 (31.7) | 61600 (22.9) | 97200 (18.7) | 73000 (56.8) | 115000 (9.2) | 93100 (33.8) | 79100 (38.7) | 83200 (22.8) | 76000 (52.2) | 93200 (13.7) | 115000 (11.7) | 94100 (7.1) | 94600 (17.3)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 2 | 0 | 2 | 0 | 2 | 1 | 0 | 2 | 18
  Cycle 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 156000 (NA) — NA = %GCV values were not reported when n<2. | 54700 (NA) — NA = %GCV values were not reported when n<2. | 57000 (NA) — NA = %GCV values were not reported when n<2. | 105000 (17.2) | 96500 (31.6) | 125000 (7.9) |  | 83500 (57.6) |  | 90800 (47.7) | 143000 (NA) — NA = %GCV values were not reported when n<2. |  | 95600 (4.66) | 97400 (23.9)

13. Secondary Outcome: Time to Maximum Concentration (Tmax) of Pembrolizumab Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 from MK-4166 plus pembrolizumab combination cohorts only and plasma isolated for analysis of pembrolizumab Tmax. Tmax was defined as time to the maximum concentration of pembrolizumab reached. Pembrolizumab Tmax was reported by dose cohort for all participants that received MK-4166 plus pembrolizumab combination therapy. Per protocol, participants receiving MK-4166 monotherapy were excluded from this analysis.
Time Frame: as for outcome 12
Population: All allocated participants who received ≥1 dose of pembrolizumab and had evaluable Tmax samples. Per protocol, MK-4166 monotherapy dose cohorts were not analyzed. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Days
  Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 2 | 3 | 3 | 4 | 23
  Cycle 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0.03 [0.03 to 0.15] | 0.06 [0.03 to 0.13] | 0.02 [0.02 to 0.03] | 0.08 [0.02 to 0.09] | 0.02 [0.02 to 0.03] | 0.03 [0.02 to 0.07] | 0.06 [0.02 to 0.13] | 0.04 [0.02 to 0.13] | 0.02 [0.02 to 0.03] | 0.11 [0.08 to 0.14] | 0.07 [0.02 to 0.13] | 0.02 [0.02 to 0.06] | 0.05 [0.02 to 0.13] | 0.02 [0.02 to 13.97]
  Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 2 | 3 | 2 | 2 | 23
  Cycle 2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0.03 [0.02 to 0.07] | 0.03 [0.03 to 0.03] | 0.03 [0.02 to 0.07] | 0.03 [0.02 to 0.13] | 0.02 [0.02 to 0.08] | 0.05 [0.03 to 0.07] | 0.03 [0.03 to 0.07] | 0.13 [0.03 to 14.1] | 0.05 [0.03 to 0.07] | 0.03 [0.02 to 0.03] | 0.06 [0.06 to 0.13] | 0.07 [0.06 to 0.08] | 0.02 [0.02 to 0.02] | 0.03 [0.02 to 1.92]
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 2 | 18
  Cycle 3 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0.03 [0.03 to 0.13] | 0.03 [0.03 to 0.03] | 0.03 [0.02 to 0.03] | 0.07 [0.02 to 0.94] | 0.02 [0.02 to 0.08] | 0.05 [0.02 to 0.08] | 0.03 [0.02 to 0.07] | 0.05 [0.03 to 0.06] | 0.05 [0.03 to 0.06] | 0.93 [0.02 to 14.16] | 0.02 [0.02 to 0.06] | 0.08 [0.02 to 0.13] | 0.10 [0.07 to 0.13] | 0.05 [0.02 to 0.13]
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 2 | 0 | 2 | 0 | 2 | 1 | 0 | 2 | 18
  Cycle 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0.13 [0.13 to 0.13] | 0.08 [0.08 to 0.08] | 0.04 [0.04 to 0.04] | 0.04 [0.02 to 0.07] | 0.04 [0.02 to 0.07] | 0.07 [0.07 to 0.07] |  | 0.03 [0.02 to 0.03] |  | 7.07 [0.02 to 14.13] | 0.10 [0.10 to 0.10] |  | 0.02 [0.02 to 0.03] | 0.03 [0.02 to 0.94]

14. Secondary Outcome: Terminal Half-Life (t ½) of Pembrolizumab Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 from MK-4166 plus pembrolizumab combination cohorts only and plasma isolated for analysis of pembrolizumab t½. t½ was defined as the time required to divide the pembrolizumab plasma concentration by two after reaching pseudo-equilibrium, following a single dose of pembrolizumab. Pembrolizumab t½ was reported by dose cohort for all participants that received MK-4166 plus pembrolizumab combination therapy. Per protocol, participants receiving MK-4166 monotherapy were excluded from this analysis.
Time Frame: as for outcome 12
Population: All allocated participants who received ≥1 dose of pembrolizumab and had evaluable t½ samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants, and MK-4166 monotherapy dose cohorts were not analyzed. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Days
  Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 2 | 2 | 3 | 4 | 22
  Cycle 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 17.2 (21.8) | 12.1 (80.3) | 14.7 (32.7) | 23.5 (54.4) | 11.8 (46.4) | 9.45 (61.8) | 10.9 (43.5) | 17.7 (23.1) | 11.3 (22.9) | 16.1 (27.6) | 13.2 (63.6) | 8.84 (189.6) | 11.2 (64.2) | 19.0 (54.1)
  Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 2 | 2 | 2 | 3 | 2 | 2 | 19
  Cycle 2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 16.8 (30.6) | 21.1 (22.4) | 10 (189.6) | 18.5 (13.4) | 14.4 (42.1) | 16.0 (4.4) | 15.0 (9.17) | 18.6 (38.1) | 12.7 (22.4) | 15.7 (9.65) | 13.7 (18.6) | 18.9 (1.03) | 17.6 (35.9) | 16.7 (55.1)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 2 | 1 | 3 | 2 | 2 | 18
  Cycle 3 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 14.0 (59.2) | 10.5 (42.1) | 14.6 (39.4) | 15.2 (49.2) | 15.0 (122.9) | 14.8 (5.7) | 9.45 (35.3) | 20.8 (15.4) | 9.38 (6.03) | 13.3 (NA) — NA = %GCV values were not reported when n<2. | 11.3 (45.2) | 8.11 (63.8) | 19.8 (11.1) | 24.9 (57.4)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 18
  Cycle 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 17.7 (NA) — NA = %GCV values were not reported when n<2. | 11.1 (NA) — NA = %GCV values were not reported when n<2. | 10.5 (NA) — NA = %GCV values were not reported when n<2. | 18.0 (117.5) | 34.1 (NA) — NA = %GCV values were not reported when n<2. | 14.9 (NA) — NA = %GCV values were not reported when n<2. |  | 23.3 (38.1) |  | 22.4 (NA) — NA = %GCV values were not reported when n<2. | 15.7 (NA) — NA = %GCV values were not reported when n<2. |  | 6.94 (34.8) | 16.6 (109.6)

15. Secondary Outcome: Area Under the Concentration-Time Curve of Pembrolizumab From Time Zero to 21 Hours After Dosing (AUC 0-21) Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 from MK-4166 plus pembrolizumab combination cohorts only and plasma isolated for analysis of pembrolizumab AUC0-21. AUC0-21 was defined as the area under the concentration-time curve of pembrolizumab from time zero to 21 hours after dosing. Pembrolizumab AUC0-21 was reported by dose cohort for all participants that received MK-4166 plus pembrolizumab combination therapy. Per protocol, participants receiving MK-4166 monotherapy were excluded from this analysis.
Time Frame: Cycles 1-4: Day 1 pre-dose, at end of pembro infusion (up to 10 minutes), at end of MK-4166 infusion (up to 10 minutes), ~2 hours after start of MK-4166 infusion, Day 2. Each cycle was 21 days. (Up to ~3 months)
Population: All allocated participants who received ≥1 dose of pembrolizumab and had evaluable AUC0-21 samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants, and MK-4166 monotherapy dose cohorts were not analyzed. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days•ng/mL
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Days•ng/mL
  Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 2 | 2 | 3 | 4 | 22
  Cycle 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 587000 (36.0) | 484000 (33.8) | 408000 (10.7) | 664000 (15.8) | 404000 (46.4) | 511000 (32.3) | 535000 (31.1) | 454000 (26.0) | 516000 (29.0) | 664000 (9.7) | 560000 (26.5) | 485000 (92.9) | 599000 (34.6) | 619000 (33.9)
  Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 2 | 2 | 2 | 3 | 2 | 2 | 19
  Cycle 2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 847000 (33.5) | 672000 (45.4) | 405000 (62.8) | 952000 (12.6) | 579000 (46.1) | 871000 (16.5) | 750000 (47.9) | 739000 (48.8) | 715000 (27.9) | 921000 (18.1) | 825000 (21.0) | 991000 (14.5) | 925000 (7.5) | 825000 (32.1)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 2 | 1 | 3 | 2 | 2 | 18
  Cycle 3 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 913000 (53.8) | 662000 (38.5) | 622000 (2.3) | 1120000 (14.1) | 633000 (59.6) | 927000 (8.1) | 738000 (37.4) | 903000 (50.6) | 752000 (27.4) | 1220000 (NA) — NA = %GCV values were not reported when n<2. | 822000 (30.2) | 883000 (25.5) | 967000 (6.3) | 1010000 (25.2)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 18
  Cycle 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1540000 (NA) — NA = %GCV values were not reported when n<2. | 490000 (NA) — NA = %GCV values were not reported when n<2. | 613000 (NA) — NA = %GCV values were not reported when n<2. | 1050000 (38.7) | 1370000 (NA) — NA = %GCV values were not reported when n<2. | 1010000 (14.7) |  | 964000 (41.8) |  | 1370000 (NA) — NA = %GCV values were not reported when n<2. | 1460000 (NA) — NA = %GCV values were not reported when n<2. |  | 810000 (27.7) | 892000 (59.3)

16. Secondary Outcome: Area Under the Concentration-Time Curve of Pembrolizumab From Time Zero to The Last Quantifiable Sample (AUC 0-last) Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 from MK-4166 plus pembrolizumab combination cohorts only and plasma isolated for analysis of pembrolizumab AUC0-last. AUC0-last was defined as the area under the concentration-time curve of pembrolizumab from time zero to the last quantifiable sample. Pembrolizumab AUC0-last was reported by dose cohort for all participants that received MK-4166 plus pembrolizumab combination therapy. Per protocol, participants receiving MK-4166 monotherapy were excluded from this analysis.
Time Frame: as for outcome 12
Population: All allocated participants who received ≥1 dose of pembrolizumab and had evaluable AUC0-last samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants, and MK-4166 monotherapy dose cohorts were not analyzed. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days•ng/mL
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Days•ng/mL
  Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 2 | 3 | 3 | 4 | 22
  Cycle 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 587000 (36.0) | 356000 (79.5) | 398000 (14.3) | 663000 (16.1) | 410000 (44.5) | 491000 (39.9) | 482000 (48.7) | 414000 (35.3) | 415000 (73.7) | 663000 (9.5) | 549000 (18.7) | 389000 (162.2) | 416000 (119.9) | 624000 (34.3)
  Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2 | 2 | 3 | 2 | 2 | 23
  Cycle 2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 847000 (33.4) | 664000 (45.0) | 321000 (125.7) | 949000 (12.7) | 573000 (47.1) | 985000 (34.7) | 759000 (47.9) | 567000 (62.3) | 766000 (18.0) | 932000 (15.8) | 873000 (14.4) | 958000 (9.49) | 1080000 (29.5) | 635000 (78.4)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 2 | 18
  Cycle 3 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 466000 (258.9) | 515000 (43.0) | 554000 (14.0) | 998000 (4.5) | 603000 (64.7) | 938000 (6.3) | 454000 (20.5) | 747000 (32.3) | 604000 (26.5) | 455000 (192.8) | 492000 (88.7) | 264000 (343.2) | 981000 (8.1) | 1080000 (33.4)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 0 | 2 | 0 | 2 | 1 | 0 | 2 | 18
  Cycle 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1550000 (NA) — NA = %GCV values were not reported when n<2. | 490000 (NA) — NA = %GCV values were not reported when n<2. | 304000 (NA) — NA = %GCV values were not reported when n<2. | 775000 (110.7) | 98800 (96422.3) | 1120000 (72.3) |  | 1020000 (33.7) |  | 1280000 (8.0) | 1410000 (NA) — NA = %GCV values were not reported when n<2. |  | 284000 (95.5) | 664000 (132.9)

17. Secondary Outcome: Area Under the Concentration-Time Curve of Pembrolizumab From Time Zero to Infinity (AUC 0-inf) Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 from MK-4166 plus pembrolizumab combination cohorts only and plasma isolated for analysis of pembrolizumab AUC0-inf. AUC0-inf was defined as the area under the concentration-time curve of pembrolizumab from time zero to infinity. Pembrolizumab AUC0-inf was reported by dose cohort for all participants that received MK-4166 plus pembrolizumab combination therapy. Per protocol, participants receiving MK-4166 monotherapy were excluded from this analysis.
Time Frame: as for outcome 12
Population: All allocated participants who received ≥1 dose of pembrolizumab and had evaluable AUC0-inf samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants, and MK-4166 monotherapy dose cohorts were not analyzed. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days•ng/mL
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Days•ng/mL
  Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 2 | 2 | 3 | 4 | 22
  Cycle 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 985000 (28.0) | 709000 (46.3) | 647000 (11.8) | 1400000 (15.6) | 582000 (65.7) | 666000 (54.4) | 740000 (39.0) | 786000 (37.5) | 703000 (36.0) | 1090000 (23.0) | 858000 (58.4) | 707000 (148.2) | 855000 (55.9) | 1130000 (68.7)
  Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 2 | 2 | 2 | 3 | 2 | 2 | 19
  Cycle 2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1450000 (51.4) | 1280000 (47.7) | 655000 (104.6) | 1700000 (21.3) | 915000 (75.1) | 1410000 (19.6) | 1210000 (50.6) | 1390000 (24.5) | 1030000 (19.3) | 1540000 (16.3) | 1260000 (23.3) | 1820000 (13.2) | 1620000 (27.2) | 1470000 (57.8)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 2 | 1 | 3 | 2 | 2 | 18
  Cycle 3 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 1440000 (94.2) | 890000 (44.1) | 1000000 (21.1) | 1870000 (36.7) | 1110000 (149.0) | 1450000 (7.0) | 949000 (37.0) | 1770000 (41.9) | 954000 (30.3) | 1870000 (NA) — NA = %GCV values were not reported when n<2. | 1160000 (56.1) | 1090000 (48.3) | 1820000 (0.2) | 2340000 (55.1)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 18
  Cycle 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 2670000 (NA) — NA = %GCV values were not reported when n<2. | 667000 (NA) — NA = %GCV values were not reported when n<2. | 816000 (NA) — NA = %GCV values were not reported when n<2. | 1980000 (118.7) | 3890000 (NA) — NA = %GCV values were not reported when n<2. | 1430000 (NA) — NA = %GCV values were not reported when n<2. |  | 2070000 (71.7) |  | 2710000 (NA) — NA = %GCV values were not reported when n<2. | 2440000 (NA) — NA = %GCV values were not reported when n<2. |  | 931000 (38.4) | 1730000 (112.9)

18. Secondary Outcome: Apparent Clearance (CL) of Pembrolizumab Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 from MK-4166 plus pembrolizumab combination cohorts only and plasma isolated for analysis of pembrolizumab CL. CL was defined as the volume of plasma from which pembrolizumab is eliminated per unit time following IV pembrolizumab administration. Pembrolizumab CL was reported by dose cohort for all participants that received MK-4166 plus pembrolizumab combination therapy. Per protocol, participants receiving MK-4166 monotherapy were excluded from this analysis.
Time Frame: as for outcome 12
Population: All allocated participants who received ≥1 dose of pembrolizumab and had evaluable CL samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants, and MK-4166 monotherapy dose cohorts were not analyzed. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/Day
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
L/Day
  Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 2 | 2 | 3 | 4 | 22
  Cycle 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0.203 (28.0) | 0.282 (46.3) | 0.309 (11.8) | 0.143 (15.6) | 0.344 (65.7) | 0.301 (54.4) | 0.270 (39.0) | 0.255 (37.6) | 0.284 (36.0) | 0.184 (22.9) | 0.233 (58.3) | 0.283 (148.4) | 0.234 (55.9) | 0.176 (68.7)
  Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 2 | 2 | 2 | 3 | 2 | 2 | 19
  Cycle 2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0.236 (33.5) | 0.298 (45.4) | 0.494 (62.7) | 0.210 (12.6) | 0.346 (46.1) | 0.230 (16.5) | 0.267 (47.9) | 0.271 (48.9) | 0.280 (27.9) | 0.217 (18.1) | 0.242 (20.9) | 0.202 (14.5) | 0.216 (7.5) | 0.242 (32.1)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 2 | 1 | 3 | 2 | 2 | 18
  Cycle 3 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0.219 (53.8) | 0.302 (38.5) | 0.322 (2.3) | 0.178 (14.1) | 0.316 (59.5) | 0.216 (8.1) | 0.271 (37.4) | 0.222 (50.7) | 0.266 (27.4) | 0.164 (NA) — NA = %GCV values were not reported when n<2. | 0.243 (30.1) | 0.227 (25.5) | 0.207 (6.3) | 0.199 (25.2)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 18
  Cycle 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 0.130 (NA) — NA = %GCV values were not reported when n<2. | 0.408 (NA) — NA = %GCV values were not reported when n<2. | 0.326 (NA) — NA = %GCV values were not reported when n<2. | 0.190 (38.6) | 0.146 (NA) — NA = %GCV values were not reported when n<2. | 0.198 (14.7) |  | 0.207 (41.9) |  | 0.147 (NA) — NA = %GCV values were not reported when n<2. | 0.137 (NA) — NA = %GCV values were not reported when n<2. |  | 0.247 (27.7) | 0.224 (59.3)

19. Secondary Outcome: Apparent Volume of Distribution (V) of Pembrolizumab Over Time
Description: Blood samples were collected at pre-specified time points during Cycles 1-4 from MK-4166 plus pembrolizumab combination cohorts only and plasma isolated for analysis of pembrolizumab V. V was defined as the theoretical volume that would be necessary to contain the total amount of administered pembrolizumab at the same concentration that it is observed in the blood plasma. Pembrolizumab V was reported by dose cohort for all participants that received MK-4166 plus pembrolizumab combination therapy. Per protocol, participants receiving MK-4166 monotherapy were excluded from this analysis.
Time Frame: as for outcome 12
Population: All allocated participants who received ≥1 dose of pembrolizumab and had evaluable V samples. Per protocol, %GCV values were not reported for cohorts with n<2 participants, and MK-4166 monotherapy dose cohorts were not analyzed. Participants with samples that were hemolyzed or analyzed outside of stability were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 4 | 23
Liters
  Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 3 | 3 | 3 | 4 | 3 | 3 | 2 | 2 | 3 | 4 | 22
  Cycle 1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 5.03 (46.6) | 4.92 (60.7) | 6.55 (21.6) | 4.85 (37.3) | 5.84 (28.1) | 4.10 (6.1) | 4.25 (37.9) | 6.50 (19.5) | 4.62 (23.8) | 4.27 (4.5) | 4.43 (4.2) | 3.61 (30.0) | 3.78 (16.7) | 4.84 (32.3)
  Cycle 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 2 | 2 | 2 | 3 | 2 | 2 | 19
  Cycle 2 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 5.52 (17.2) | 8.13 (53.3) | 7.76 (54.5) | 5.29 (9.3) | 6.82 (32.9) | 4.92 (11.1) | 5.70 (44.1) | 7.34 (92.9) | 4.88 (41.7) | 4.96 (20.0) | 4.71 (23.3) | 5.36 (16.6) | 5.24 (22.5) | 5.79 (38.6)
  Cycle 3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 2 | 3 | 3 | 2 | 3 | 2 | 2 | 1 | 3 | 2 | 2 | 18
  Cycle 3 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 4.31 (10.4) | 4.40 (50.6) | 6.81 (44.4) | 3.94 (39.5) | 6.73 (53.6) | 4.40 (7.7) | 3.62 (55.0) | 6.51 (62.6) | 3.63 (20.5) | 3.24 (NA) — NA = %GCV values were not reported when n<2. | 4.01 (15.4) | 2.64 (33.9) | 5.66 (14.9) | 7.09 (73.6)
  Cycle 4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 18
  Cycle 4 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 3.10 (NA) — NA = %GCV values were not reported when n<2. | 6.37 (NA) — NA = %GCV values were not reported when n<2. | 4.92 (NA) — NA = %GCV values were not reported when n<2. | 4.78 (54.9) | 7.05 (NA) — NA = %GCV values were not reported when n<2. | 4.47 (NA) — NA = %GCV values were not reported when n<2. |  | 6.85 (6.4) |  | 4.31 (NA) — NA = %GCV values were not reported when n<2. | 3.17 (NA) — NA = %GCV values were not reported when n<2. |  | 2.46 (7.2) | 5.48 (44.7)

20. Secondary Outcome: Glucocorticoid-Induced Tumor Necrosis Factor Receptor-Related Protein (GITR) Receptor Availability Following MK-4166 Administration
Description: GITR protein receptor is internalized upon binding by MK-4166. To evaluate GITR target engagement, a GITR receptor availability assay was developed to assess the availability of cell surface GITR following administration of MK-4166. GITR was detected on CD4+CD25+ and CD4+CD95+ T-cell sub-populations in peripheral blood using flow cytometry. GITR receptor availability on representative CD4+ CD25+ T cell subsets following MK-4166 administration was reported over time for each dose cohort.
Time Frame: Cycle 1 Day 1: at end of infusion (up to 10 minutes), 2 hours post-infusion, Cycle 1 Days 2, 3, 5, 8, 15, Cycle 2 Day 1 pre-dose. Each cycle was 21 days.
Population: All allocated participants who received at least 1 dose of MK-4166 and had evaluable flow cytometry data.
Measure: Mean (Standard Deviation); unit: Percentage GITR receptor availability
Groups:
- MK-4166 3.3 mg: Participants received 3.3 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
- MK-4166 670 mg: Participant received 670 mg MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles.
Arm/Group | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
Number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 5 | 3 | 3 | 3 | 3 | 3 | 5 | 3 | 3 | 1 | 3 | 3 | 4 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 20
Percentage GITR receptor availability
  Cycle 1:Day 1; End of Infusion: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 5 | 3 | 3 | 3 | 2 | 3 | 4 | 3 | 3 | 1 | 3 | 3 | 4 | 3 | 2 | 3 | 3 | 3 | 0 | 3 | 3 | 3 | 3 | 3 | 20
  Cycle 1:Day 1; End of Infusion | 103.7 (NA) — NA = SD values were not reported when n<2. |  | 52.8 (NA) — NA = SD values were not reported when n<2. | 92.5 (NA) — NA = SD values were not reported when n<2. | 51.9 (NA) — NA = SD values were not reported when n<2. | 8.8 (NA) — NA = SD values were not reported when n<2. | 4.6 (NA) — NA = SD values were not reported when n<2. |  | 3.0 (NA) — NA = SD values were not reported when n<2. | 26.3 (32.0) | 10.8 (9.9) | 9.1 (3.2) | 4.2 (2.7) | 41.9 (4.7) | 7.4 (5.9) | 9.5 (6.5) | 13.9 (3.4) | 15.0 (9.8) | 26.0 (NA) — NA = SD values were not reported when n<2. | 14.4 (15.1) | 6.9 (3.2) | 4.2 (1.5) | 7.3 (3.6) | 7.6 (6.8) | 7.0 (2.6) | 4.6 (2.3) | 19.9 (15.4) |  | 46.5 (54.5) | 8.8 (5.3) | 26.8 (18.4) | 28.4 (28.3) | 10.5 (8.9) | 13.3 (17.4)
  Cycle 1:Day 1; 2 hours Post Infusion: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1:Day 1; 2 hours Post Infusion | 102.5 (NA) — NA = SD values were not reported when n<2. |  | 63.2 (NA) — NA = SD values were not reported when n<2. | 91.7 (NA) — NA = SD values were not reported when n<2. | 42.7 (NA) — NA = SD values were not reported when n<2. | 17.0 (NA) — NA = SD values were not reported when n<2. | 2.4 (NA) — NA = SD values were not reported when n<2. |  | 1.2 (NA) — NA = SD values were not reported when n<2. | 0.7 (NA) — NA = SD values were not reported when n<2. |  | 6.9 (NA) — NA = SD values were not reported when n<2. |  |  |  |  |  |  |  |  | 4.9 (2.5) | 3.0 (2.1) | 8.1 (4.8) | 9.1 (NA) — NA = SD values were not reported when n<2. |  |  |  |  |  |  |  |  |  |
  Cycle 1: Day 2: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 5 | 2 | 3 | 3 | 3 | 3 | 5 | 3 | 3 | 1 | 3 | 3 | 4 | 2 | 3 | 2 | 3 | 2 | 0 | 2 | 3 | 2 | 3 | 1 | 20
  Cycle 1: Day 2 | 107.0 (NA) — NA = SD values were not reported when n<2. |  | 59.5 (NA) — NA = SD values were not reported when n<2. | 96.9 (NA) — NA = SD values were not reported when n<2. | 55.4 (NA) — NA = SD values were not reported when n<2. | 9.5 (NA) — NA = SD values were not reported when n<2. | 2.2 (NA) — NA = SD values were not reported when n<2. |  | 3.3 (NA) — NA = SD values were not reported when n<2. | 46.2 (86.4) | 15.2 (3.0) | 4.8 (1.0) | 17.4 (24.6) | 30.4 (34.6) | 5.8 (5.2) | 14.7 (7.1) | 12.0 (8.9) | 6.7 (2.6) | 82.5 (NA) — NA = SD values were not reported when n<2. | 20.0 (10.7) | 6.1 (3.1) | 2.4 (0.3) | 7.3 (4.0) | 7.1 (1.2) | 6.5 (0.2) | 7.4 (2.2) | 6.7 (4.6) |  | 5.9 (0.9) | 11.4 (4.2) | 23.0 (3.4) | 26.0 (32.2) | 13.7 (NA) — NA = SD values were not reported when n<2. | 15.6 (20.8)
  Cycle 1: Day 3: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Cycle 1: Day 3 | 109.1 (NA) — NA = SD values were not reported when n<2. |  | 108.3 (NA) — NA = SD values were not reported when n<2. | 85.4 (NA) — NA = SD values were not reported when n<2. | 72.4 (NA) — NA = SD values were not reported when n<2. | 5.4 (NA) — NA = SD values were not reported when n<2. | 2.6 (NA) — NA = SD values were not reported when n<2. |  | 0.9 (NA) — NA = SD values were not reported when n<2. | 50.0 (70.1) |  | 4.3 (NA) — NA = SD values were not reported when n<2. |  |  |  |  |  |  |  |  | 7.2 (3.5) | 2.4 (1.3) | 3.9 (1.3) | 1.6 (NA) — NA = SD values were not reported when n<2. |  |  |  |  |  |  |  | 9.9 (NA) — NA = SD values were not reported when n<2. |  |
  Cycle 1: Day 5: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 1: Day 5 | 97.5 (NA) — NA = SD values were not reported when n<2. |  | 107.1 (NA) — NA = SD values were not reported when n<2. | 111.6 (NA) — NA = SD values were not reported when n<2. | 83.0 (NA) — NA = SD values were not reported when n<2. | 8.8 (NA) — NA = SD values were not reported when n<2. | 1.7 (NA) — NA = SD values were not reported when n<2. |  | 4.5 (NA) — NA = SD values were not reported when n<2. |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |
  Cycle 1: Day 8: number analyzed (Participants) | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 5 | 3 | 3 | 3 | 2 | 3 | 4 | 3 | 3 | 1 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 1 | 1 | 3 | 2 | 2 | 1 | 18
  Cycle 1: Day 8 | 100.2 (NA) — NA = SD values were not reported when n<2. |  | 103.4 (NA) — NA = SD values were not reported when n<2. | 114.9 (NA) — NA = SD values were not reported when n<2. | 89.2 (NA) — NA = SD values were not reported when n<2. | 15.0 (NA) — NA = SD values were not reported when n<2. | 8.2 (NA) — NA = SD values were not reported when n<2. |  |  | 148.6 (281.6) | 5.8 (4.3) | 6.3 (5.1) | 10.0 (8.3) | 10.2 (3.6) | 2.2 (0.4) | 16.0 (9.4) | 19.3 (15.3) | 22.5 (12.6) | 82.9 (NA) — NA = SD values were not reported when n<2. | 15.5 (11.3) | 10.2 (8.9) | 2.9 (2.3) | 5.4 (4.6) | 12.8 (7.1) | 3.8 (1.8) | 6.0 (4.9) | 9.3 (4.9) | 8.6 (NA) — NA = SD values were not reported when n<2. | 4.0 (NA) — NA = SD values were not reported when n<2. | 11.8 (7.0) | 12.0 (5.6) | 25.3 (3.0) | 8.8 (NA) — NA = SD values were not reported when n<2. | 11.3 (13.1)
  Cycle 1: Day 15: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 5 | 2 | 1 | 2 | 1 | 3 | 3 | 3 | 2 | 1 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 1 | 1 | 1 | 3 | 3 | 2 | 2 | 18
  Cycle 1: Day 15 |  |  | 123.9 (NA) — NA = SD values were not reported when n<2. | 122.9 (NA) — NA = SD values were not reported when n<2. | 94.8 (NA) — NA = SD values were not reported when n<2. | 74.8 (NA) — NA = SD values were not reported when n<2. | 71.4 (NA) — NA = SD values were not reported when n<2. |  | 71.2 (NA) — NA = SD values were not reported when n<2. | 169.3 (301.5) | 2.2 (1.6) | 4.0 (NA) — NA = SD values were not reported when n<2. | 40.9 (28.1) | 6.5 (NA) — NA = SD values were not reported when n<2. | 8.9 (13.8) | 15.2 (15.9) | 8.1 (6.7) | 4.8 (2.7) | 65.8 (NA) — NA = SD values were not reported when n<2. | 15.5 (5.6) | 39.9 (49.1) | 4.8 (1.8) | 8.8 (9.2) | 11.4 (8.7) | 5.0 (4.3) | 9.1 (4.8) | 28.6 (NA) — NA = SD values were not reported when n<2. | 12.5 (NA) — NA = SD values were not reported when n<2. | 22.2 (NA) — NA = SD values were not reported when n<2. | 3.8 (1.5) | 40.8 (54.4) | 22.5 (8.7) | 21.9 (17.6) | 13.0 (14.0)
  Cycle 2: Day 1; Pre-dose: number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 3 | 2 | 2 | 3 | 3 | 2 | 3 | 2 | 3 | 1 | 3 | 3 | 3 | 3 | 2 | 2 | 1 | 1 | 2 | 2 | 3 | 3 | 2 | 2 | 18
  Cycle 2: Day 1; Pre-dose | 106.0 (NA) — NA = SD values were not reported when n<2. |  |  | 114.9 (NA) — NA = SD values were not reported when n<2. | 92.2 (NA) — NA = SD values were not reported when n<2. | 80.3 (NA) — NA = SD values were not reported when n<2. |  |  | 84.8 (NA) — NA = SD values were not reported when n<2. | 49.3 (84.6) | 57.1 (52.9) | 67.4 (91.5) | 7.6 (5.5) | 7.8 (3.8) | 29.3 (28.1) | 44.8 (62.4) | 17.7 (5.7) | 39.0 (50.0) | 77.0 (NA) — NA = SD values were not reported when n<2. | 7.0 (3.6) | 109.9 (37.2) | 74.1 (36.4) | 70.0 (51.8) | 11.7 (7.9) | 12.6 (6.9) | 13.5 (NA) — NA = SD values were not reported when n<2. | 51.2 (NA) — NA = SD values were not reported when n<2. | 8.3 (5.8) | 7.3 (9.3) | 13.0 (12.5) | 55.5 (43.2) | 8.0 (7.8) | 27.4 (19.2) | 9.2 (9.4)

ADVERSE EVENTS:
Time Frame: Up to approximately 61 months (through final cut-off date of 31-Jul-2019)
Description: All-Cause Mortality table includes all allocated participants.
  Serious and Other adverse events (AEs) include all allocated participants who received ≥1 dose of study drug. Per protocol, disease progression of cancer on study not considered an AE unless considered related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs. Data reported by treatment arm and by dose cohort
Groups:
- MK-4166: All participants that received MK-4166 IV on Day 1 of each 21-day cycle, for up to 4 cycles (according to assigned dose).
- MK-4166 + Pembro: All participants that received MK-4166 IV on Day 1 of each 21-day cycle for up to 4 cycles (according to assigned dose) plus pembrolizumab 200 mg IV on Day 1 of each 21-day cycle for up to 35 cycles (according to assigned doses).
Arm/Group | MK-4166 | MK-4166 + Pembro | MK-4166 0.0015 mg | MK-4166 0.0045 mg | MK-4166 0.014 mg | MK-4166 0.04 mg | MK-4166 0.12 mg | MK-4166 0.37 mg | MK-4166 1.1 mg | MK-4166 3.3 mg | MK-4166 10 mg | MK-4166 30 mg | MK-4166 42 mg | MK-4166 59 mg | MK-4166 82 mg | MK-4166 120 mg | MK-4166 170 mg | MK-4166 240 mg | MK-4166 340 mg | MK-4166 480 mg | MK-4166 670 mg | MK-4166 900 mg | MK-4166 1.1 mg + Pembro | MK-4166 3.3 mg + Pembro | MK-4166 10 mg + Pembro | MK-4166 30 mg + Pembro | MK-4166 42 mg + Pembro | MK-4166 59 mg + Pembro | MK-4166 82 mg + Pembro | MK-4166 120 mg + Pembro | MK-4166 170 mg + Pembro | MK-4166 240 mg + Pembro | MK-4166 340 mg + Pembro | MK-4166 480 mg + Pembro | MK-4166 670 mg + Pembro | MK-4166 900 mg + Pembro
All-Cause Mortality (participants affected / at risk) | 16/50 | 13/66 | 0/1 | 1/1 | 1/1 | 0/1 | 0/1 | 0/1 | 0/1 | 1/1 | 0/1 | 3/6 | 0/3 | 1/3 | 0/4 | 1/3 | 1/3 | 2/5 | 1/4 | 1/3 | 1/3 | 2/4 | 0/3 | 1/5 | 1/3 | 0/3 | 0/3 | 2/3 | 2/4 | 0/3 | 0/3 | 0/3 | 1/3 | 1/3 | 2/4 | 3/23
Serious Adverse Events (participants affected / at risk) | 6/48 | 21/65 | 0/1 | 1/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 2/6 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/5 | 1/4 | 2/3 | 0/3 | 0/3 | 1/3 | 1/4 | 1/3 | 0/3 | 2/3 | 3/3 | 1/4 | 0/3 | 0/3 | 1/3 | 1/3 | 1/3 | 2/4 | 7/23
Other Adverse Events (participants affected / at risk) | 43/48 | 63/65 | 0/1 | 1/1 | 1/1 | 1/1 | 1/1 | 1/1 | 1/1 | 1/1 | 1/1 | 4/6 | 3/3 | 3/3 | 2/3 | 2/3 | 3/3 | 5/5 | 4/4 | 3/3 | 3/3 | 3/3 | 3/3 | 3/4 | 3/3 | 3/3 | 3/3 | 3/3 | 4/4 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 4/4 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-4166 (N=48) | MK-4166 + Pembro (N=65) | MK-4166 0.0015 mg (N=1) | MK-4166 0.0045 mg (N=1) | MK-4166 0.014 mg (N=1) | MK-4166 0.04 mg (N=1) | MK-4166 0.12 mg (N=1) | MK-4166 0.37 mg (N=1) | MK-4166 1.1 mg (N=1) | MK-4166 3.3 mg (N=1) | MK-4166 10 mg (N=1) | MK-4166 30 mg (N=6) | MK-4166 42 mg (N=3) | MK-4166 59 mg (N=3) | MK-4166 82 mg (N=3) | MK-4166 120 mg (N=3) | MK-4166 170 mg (N=3) | MK-4166 240 mg (N=5) | MK-4166 340 mg (N=4) | MK-4166 480 mg (N=3) | MK-4166 670 mg (N=3) | MK-4166 900 mg (N=3) | MK-4166 1.1 mg + Pembro (N=3) | MK-4166 3.3 mg + Pembro (N=4) | MK-4166 10 mg + Pembro (N=3) | MK-4166 30 mg + Pembro (N=3) | MK-4166 42 mg + Pembro (N=3) | MK-4166 59 mg + Pembro (N=3) | MK-4166 82 mg + Pembro (N=4) | MK-4166 120 mg + Pembro (N=3) | MK-4166 170 mg + Pembro (N=3) | MK-4166 240 mg + Pembro (N=3) | MK-4166 340 mg + Pembro (N=3) | MK-4166 480 mg + Pembro (N=3) | MK-4166 670 mg + Pembro (N=4) | MK-4166 900 mg + Pembro (N=23)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-4166 (N=48) | MK-4166 + Pembro (N=65) | MK-4166 0.0015 mg (N=1) | MK-4166 0.0045 mg (N=1) | MK-4166 0.014 mg (N=1) | MK-4166 0.04 mg (N=1) | MK-4166 0.12 mg (N=1) | MK-4166 0.37 mg (N=1) | MK-4166 1.1 mg (N=1) | MK-4166 3.3 mg (N=1) | MK-4166 10 mg (N=1) | MK-4166 30 mg (N=6) | MK-4166 42 mg (N=3) | MK-4166 59 mg (N=3) | MK-4166 82 mg (N=3) | MK-4166 120 mg (N=3) | MK-4166 170 mg (N=3) | MK-4166 240 mg (N=5) | MK-4166 340 mg (N=4) | MK-4166 480 mg (N=3) | MK-4166 670 mg (N=3) | MK-4166 900 mg (N=3) | MK-4166 1.1 mg + Pembro (N=3) | MK-4166 3.3 mg + Pembro (N=4) | MK-4166 10 mg + Pembro (N=3) | MK-4166 30 mg + Pembro (N=3) | MK-4166 42 mg + Pembro (N=3) | MK-4166 59 mg + Pembro (N=3) | MK-4166 82 mg + Pembro (N=4) | MK-4166 120 mg + Pembro (N=3) | MK-4166 170 mg + Pembro (N=3) | MK-4166 240 mg + Pembro (N=3) | MK-4166 340 mg + Pembro (N=3) | MK-4166 480 mg + Pembro (N=3) | MK-4166 670 mg + Pembro (N=4) | MK-4166 900 mg + Pembro (N=23)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 12 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 11 (13) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Ascites (Gastrointestinal disorders) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (7) | 8 (9) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 9 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (10) | 16 (17) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (10) | 13 (18) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (6)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site scar (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chills (General disorders) | 2 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 15 (15) | 37 (42) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 14 (17)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (6) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Oral candidiasis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Urinary tract infection (Infections and infestations) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 9 (13) | 22 (27) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 3 (3) | 10 (13)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 12 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 9 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 5 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 13 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 6 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmetria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal rash (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 11 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (9) | 15 (18) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contrast media reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menopause (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT02132754/Prot_SAP_000.pdf